CLINICAL TRIAL: NCT01677715
Title: Study on Evaluating the Promote Effect of Yili Mei Yi Tian Active Lactobacillus Drink on Immunity and Physical Intestinal Canal
Brief Title: Study of Yili Mei Yi Tian Active Lactobacillus Drink to Improve Immunity and Digestive System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Yili Industrial Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YL/CL-003
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Immunization; Human Influenza; Common Cold; Constipation; Dyspepsia; Flatulence; Abdominal Pain
MeSH Terms: conditions — Influenza, Human; Common Cold; Constipation; Dyspepsia; Flatulence; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Yili "Mei Yi Tian" lactobacillus drink (Active Comparator): 100ml of Yili "Mei Yi Tian" active lactobacillus drink to be taken once per day at 10am daily during the 84-days intervention
  Interventions: Dietary Supplement: Yili "Mei Yi Tian" active lactobacillus drink
- recombined milk drink contains no lactobacillus (Placebo Comparator): 100ml of recombined milk drink contains no lactobacillus to be taken once per day at 10am daily during the 84-days intervention
  Interventions: Dietary Supplement: recombined milk drink contains no lactobacillus

INTERVENTIONS:
Dietary Supplement: Yili "Mei Yi Tian" active lactobacillus drink — 100ml of Yili "Mei Yi Tian" active lactobacillus drink to be taken once per day at 10am daily during the 84-days intervention
  Arms: Yili "Mei Yi Tian" lactobacillus drink
Dietary Supplement: recombined milk drink contains no lactobacillus — 100ml of recombined milk drink contains no lactobacillus to be taken once per day at 10am daily during the 84-days intervention
  Arms: recombined milk drink contains no lactobacillus

SUMMARY:
Study on Evaluating the Promote Effect of Yili Mei Yi Tian Active Lactobacillus Drink on Immunity and Physical Intestinal Canal

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 45 years sub-health white-collars, catch cold for 4 to 6 times in last year, with low immunity;
* Non-specific and/or moderate constipation;
* Irregular or occasional gastrointestinal disorders (flatulence, gurgling, feeling heavy after eating, abdominal pain);
* Slow transit or irregular bowels movements (abnormal feces solidity, bowel movements decreased, e.g. every 2-3 days or less than 3 times per week);
* Able to understand the nature and purpose of the study including potential risks and side effects;
* Willing to consent to study participation and to comply with study requirements

Exclusion Criteria:

* Diagnosed as immunity-low associated with chronic disease;
* Diagnosed as chronic constipation;
* Treated gastrointestinal symptoms;
* Currently suffering from diarrhea;
* Suffering from rhinitis chronic, laryngitis, labored breathing that similar to flu symptoms. Such as chronic allergic rhinitis, asthma, COPD;
* Treatment by analgesic such as aspirin and paracetamol;
* Had laxatives or other remedies to promote digestion 2 weeks prior to the study start;
* Consuming dairy products or supplements containing pro/pre-biotic 10 days prior to the study start;
* Long-term use of any prescription or OTC medication that inhibit or prevent flu symptoms, including but not limited to, antihistamine, pectoral, high doses of vitamin C;
* Recent use (within 3 months of screening) of any prescription or OTC medication that significantly affects immune response, such as antibiotic;
* Recent inoculation (within 6 months of screening) of influenza vaccine, or other vaccine in 15 days;
* History of alcohol, drug, or medication abuse;
* Pregnant or breastfeeding women;
* Participation in another study with any investigational product within 3 months of screening
* Any comorbidity that could, in the opinion of the investigator, preclude the subject's ability to successfully and safely complete the study or that may confound study outcomes

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in constipation condition | Baseline & 3 months
Assess severity of flu symptoms | 3 months

SECONDARY OUTCOMES:
Change in immune markers such as antibodies and interleukins | Baseline & 3 months
Change in gut resident flora | Baseline & 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ying An, Ph.D, Study Director — Inner Mongolia Hilo Industrial Group Co., Ltd; Leiming Xu, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Digestive system Dept.; Gengru Jiang, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Kidney Dept.
Locations (2):
- China (2):
  - NanMoFang Community Health Service Center, ChaoYang District, Beijing Municipality
  - Shanghai Municipal Food and Drug Administration Baoshan Office, Baoshan District, Shanghai Municipality